CLINICAL TRIAL: NCT03630822
Title: Experimentation of a Protocol of Psychiatric Advance Directives: Randomized Controlled Multi-site Trial
Brief Title: Multicenter, Randomized, Comparative and Prospective Study Evaluating the Impact on the Care Path of an Editorial Program Accompanied by Advance Directives in Psychiatry (DAP) for People Suffering From Schizophrenia, Bipolar I Disorder or Schizoaffective Disorder
Acronym: DAiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-04; 2018-A00146-49 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia; Bipolar I Disorder
MeSH Terms: conditions — Schizophrenia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beneficiary of the advance directive program (Experimental)
  Interventions: Behavioral: Psychiatric Advanced Directive
- beneficiary of standard Support (Active Comparator)
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Psychiatric Advanced Directive — The patient completes a questionnaire to express in advance his wishes regarding his future care in psychiatry.
  Arms: beneficiary of the advance directive program
Behavioral: Standard care — standardized maintenance with the patient
  Arms: beneficiary of standard Support

SUMMARY:
Severe mental illness is accompanied by cognitive fluctuations that can alter decision-making skills and lead to coerced care. Taking into account, on the one hand, the health, social and economic impact of forced hospitalization, on the other hand the importance of self-determination, the reinforcement of the power to act in the evolution of these disorders, new strategies to better reflect the views of people have been developed.

Among these, the drafting of Advanced Directives in Psychiatric (ADP), allows people with mental disorders to write while their decision-making skills are restored care instructions in case of decompensation.

It is a tool of "advanced therapeutic education" and early prevention of relapses.

It is hypothesized that the implementation of drafting accompanied by advance directives to people with severe psychiatric disorders decreases in the short term the number of forced hospitalization care pathway of these people, compared to the subjects having not benefited from this device.

This research will take the form of a randomized controlled trial on 3 sites. The "quantitative" evaluation component of results and processes will be completed with a qualitative anthropological and socio-political evaluation component documenting the trajectories of individuals and the implementation of the program, as well as a "participatory research" component aimed at a dialogue between users, researchers and professionals.

The patient who is a beneficiary of the "Advanced Directives in Psychiatric" program will be encouraged to complete the " Advanced Directives in Psychiatric" document and will receive support in drafting them. The non-beneficiary patient of the program will follow up with his psychiatrist unchanged.

The experimental design of the quantitative component is based on an experimental, randomized, prospective, controlled, parallel study, comparing two groups of subjects with severe psychiatric disorders.

This research will assess the effectiveness, efficiency and impact of the " Advanced Directives in Psychiatric" program compared to conventional psychiatric care alone.

Ultimately, the objective of describing the effects of the program on health organizations and on the representations and practices of professionals, caregivers and users is at the service of a better understanding of the conditions of possibility of the generalization of this experimentation.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old;
* diagnosed with schizophrenia, bipolar I disorder, or schizoaffective disorder
* receiving ambulatory care by a treating psychiatrist, investigator
* having been hospitalized under duress at least once during the year preceding the inclusion
* being in decision-making jurisdiction
* can be under curator
* agreeing to participate in the study and with informed consent signed by the subject, as well as by the legal representative in the case of a person under guardianship.

Exclusion Criteria:

* less than 18 years old;
* participating in another study simultaneously
* in situations of decision-making incompetence
* not able to read and write
* refusing to participate in the study, or the legal representative refusing to participate in the study in the case of a person under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Rate of patients with compulsory admission | 12 months
  Evaluation of the hospitalization rate by comparing the two groups

SECONDARY OUTCOMES:
Evaluation of patient recovery rates | 12 months
  The rate is assessed by the Recovery Assessment Scale (RAS)
Evaluation of the empowerment rate | 12 months
  The rate is assessed by the Empowerment Scale (ES)
Measuring the health-related quality of life of patients | 12 months
  Health-related quality of life is measured using a specific scale: the S-QOL. It is a self-reported instrument of 41 items that assesses the quality of life in patients with schizophrenia
Measuring mental health symptoms of patients | 12 months
  Mental health symptoms are measured by Modified Colorado Symptom Index (MCSI)
Evaluation of the therapeutic alliance between the patient and his psychiatrist | 12 months
  The therapeutic alliance between the patient and his psychiatrist is assessed by the 4-Point Alliance Self Report (4-PAS) questionnaire
Measuring Disease Awareness | 12 months
  Disease Awareness is assessed by the évaluée par l'échelle SUMD (Scale to Assess Unawareness in Mental Disorder
Evaluation of the severity of the psychiatric disorder by the psychiatrist | 12 months
  The severity of the psychiatric disorder is assessed by the Clinical Global Impression (ICG) scale
Medico-economic analysis (cost-utility) | 12 months
  Number of inpatient
Medico-economic analysis (cost-utility) | 12 months
  Number of emergency department visits
Medico-economic analysis (cost-utility) | 12 months
  Number of outpatient visits
Medico-economic analysis (cost-utility) | 12 months
  Loss of productivity

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tinland A, Loubiere S, Mougeot F, Jouet E, Pontier M, Baumstarck K, Loundou A, Franck N, Lancon C, Auquier P; DAiP Group. Effect of Psychiatric Advance Directives Facilitated by Peer Workers on Compulsory Admission Among People With Mental Illness: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Aug 1;79(8):752-759. doi: 10.1001/jamapsychiatry.2022.1627. PMID 35662314
- [Derived] Tinland A, Leclerc L, Loubiere S, Mougeot F, Greacen T, Pontier M, Franck N, Lancon C, Boucekine M, Auquier P. Psychiatric advance directives for people living with schizophrenia, bipolar I disorders, or schizoaffective disorders: Study protocol for a randomized controlled trial - DAiP study. BMC Psychiatry. 2019 Dec 27;19(1):422. doi: 10.1186/s12888-019-2416-9. PMID 31881954